CLINICAL TRIAL: NCT01285336
Title: The Genetic and the Functional Study of DNA Repair System and the Susceptibility to Rheumatoid Arthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chung-Ming Huang, China Medical University Hospital
Purpose: Health Services Research
Other Study IDs: DMR98-IRB-309-1; NSC99-2314-B-039-005-MY3 (Other: NSC)
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2012-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis (RA); DNA repair system; polymorphism; susceptibility; copy number variation (CNV)
MeSH Terms: conditions — Arthritis, Rheumatoid; Disease Susceptibility

ARMS (1):
- The genetic and the functional study (Experimental)

INTERVENTIONS:
Genetic:

SUMMARY:
This study is valuable for the understanding the role of DNA repair system plays in the progression of rheumatoid arthritis and for the development of new therapeutic modality in the future.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a symmetric polyarticular arthritis that primarily affects the small diarthrodial joints of the hands and feet. In addition to inflammation in the synovium, which is the joint lining, the aggressive front of tissue called pannus invades and destroys local articular structures. The synovium is normally a relatively acellular structure with a delicate intimal lining. RA is also a chronic autoimmune disease and can lead to deformities and severe disabilities, due to irreversible damage of tendons, joints, and bones. It is known that RA can be considered as a complex genetic disease and many "disease-risk" genes or "disease-protective" genes can be involved. Numerous studies reported the association of IL-6, IL-8 genes with systemic lupus erythematosus (SLE) and the association of HLA-DR gene polymorphisms with RA. In addition, the chronic inflammatory process of RA is mediated through cytokines network, which leads to induce some destructive enzymes, like matrix metalloprotieases, in the cellular synovial tissue of joints. Although RA is a common arthritis with a prevalence of 1% in Taiwan, the pathogenesis is still incompletely studied, especially in DNA repair relative genes.

In this proposal, we would like to perform the following experiments:

1. Study the associations of the polymorphisms of DNA repair relative genes and the susceptibility to RA;
2. Study the associations of the copy number variation (CNV) of DNA repair relative genes and the susceptibility to RA;
3. Functional assay in DNA repair relative genes and compare it with the copy number variation (CNV), genotype and/or haplotype in RA patients; So far, we have analyzed the association between RA and several SNPs of MUTYH in DNA repair systems. We also analyzed the relationship between the SNPs results and RA using the pathological features. These data are helpful to clarify the susceptibility of RA patients with the genotype and/or haplotype in DNA repair system.

This study is valuable for the understanding the role of DNA repair system plays in the progression of rheumatoid arthritis and for the development of new therapeutic modality in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant has sang a consent form.

Exclusion Criteria:

* Participant is under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2010-08

CONTACTS AND LOCATIONS:
Locations (1):
- The Institutional Review Board China Medical University Hospital, Taichung, Taiwan